CLINICAL TRIAL: NCT06878586
Title: Diagnostic Evaluation of Esophageal Motility Disorders Using the Chicago IV Protocol in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abdelrahman Rashid abdelrhman, residant doctor, Assiut University
Other Study IDs: Esophageal Motility Chicago IV
Record Dates: First submitted 2025-03-07; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Esophageal Motility Disorders
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Adult patients (age ≥ 18 years) at Ain Shams University presenting symptoms such as dysphagia, chest pain, regurgitation, or heartburn.

SUMMARY:
Esophageal motility disorders (EMDs) encompass a spectrum of conditions characterized by abnormal movement and coordination of the esophagus, leading to symptoms such as dysphagia, chest pain, regurgitation, and heartburn . These symptoms can severely impact quality of life, often requiring detailed diagnostic evaluations for appropriate management . High-resolution esophageal manometry (HRM) has emerged as a critical diagnostic tool, providing comprehensive assessments of esophageal motility and improving our understanding of the pathophysiology behind EMDs . The advancements in HRM technology have significantly enhanced diagnostic accuracy, leading to more effective treatment strategies.

The Chicago Classification (CC) was introduced to standardize the interpretation of HRM findings and facilitate communication among clinicians. Since its inception in 2009, the classification has undergone several updates to reflect ongoing advancements. The most recent update, Chicago Classification version 4.0 (CC v4.0), resulted from two years of collaboration by an international working group of motility experts . This version places a greater emphasis on clinical relevance, refining diagnostic criteria to include standardized assessments in both the supine and upright positions, as well as the use of provocative maneuvers to provide a more thorough evaluation of esophageal function

. These enhancements aim to improve the understanding and diagnosis of complex motility disorders Although CC version 3.0 (CC v3.0) has been widely utilized, it has limitations that CC v4.0 effectively addresses to enhance esophageal motility testing. By requiring assessments in both supine and upright positions, CC v4.0 captures motility abnormalities in more physiologically relevant conditions, The inclusion of provocative testing methods, such as multiple rapid swallows (MRS) and solid swallows, further increases sensitivity for detecting disorders under stress. Moreover, CC v4.0 offers a comprehensive analysis of esophagogastric junction (EGJ) function, introducing criteria for EGJ outflow obstruction and EGJ typing, which clarify interactions with the lower esophageal sphincter . This updated framework also emphasizes bolus transit and metrics for fragmented peristalsis, facilitating the identification of subtle motility issues that may impact bolus clearance In Egypt, the majority of manometric devices are configured to automatically interpret results using CC v3.0, limiting the integration of newer diagnostic criteria. By manually applying CC v4.0 in this study, we seek to determine whether its updated metrics offer enhanced diagnostic precision and a better correlation with clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) at Ain Shams University presenting symptoms such as dysphagia, chest pain, regurgitation, or heartburn.

Exclusion Criteria:

* Patients with prior esophageal surgeries, significant structural abnormalities, or those unable to provide informed consent will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients (age ≥ 18 years) at Ain Shams University presenting symptoms such as dysphagia, chest pain, regurgitation, or heartburn.
Sampling Method: Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Chicago Classification version 4 for esophageal motility disorders (EMDs) in the Egyptian population | baseline
  Disorders of EGJ Outflow Type I Achalasia: Abnormal median IRP & 100% failed peristalsis Type II Achalasia: Abnormal median IRP, 100% failed peristalsis, & ≥20% swallows with panesophageal pressurization Type III Achalasia: Abnormal median IRP & ≥20% swallows with premature/spastic contraction and no evidence of peristalsis